CLINICAL TRIAL: NCT07220915
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of Panzyga for Prevention of Major Infection in Patients With Hypogammaglobulinemia and Autoimmune or Rheumatic Conditions Receiving Treatment With B-cell Depletion Therapy ("PROTECT")
Brief Title: Supporting Weak Immune System During Autoimmune Therapy: Testing Panzyga to Prevent Infections
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NGAM-16
Record Dates: First submitted 2025-09-30; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Hypogammaglobulinemia; Autoimmune Conditions; Rheumatic Conditions; Infections
MeSH Terms: conditions — Agammaglobulinemia; Infections | interventions — Panzyga

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Panzyga 10% (Active Comparator): Panzyga is a 10% Ig formulation for intravenous (IV) administration. The product is delivered as a ready-to-use solution in glass bottles. Patients in the Panzyga treatment arm will receive 0.4 g/kg (4 mL/kg) per single infusion every 4 weeks for up to 48 weeks (up to 13 infusions).
  In the open-label phase patients will receive Panzyga 0.4 g/kg. If 3-4 weeks after the first open-label infusion the IgG trough level falls below 7 g/L, the dose will be increased to 0.6 g/kg. Additionally, the dose may be increased to 0.6 g/kg if a patient experiences one more major infection, or ≥2 other (non-major) infections.
  Interventions: Drug: Panzyga, 10% Intravenous Solution
- Placebo (Placebo Comparator): 4 mL/kg 0.9% w/v sodium chloride solution per single IV infusion every 4 weeks for up to 48 weeks (up to 13 infusions).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Panzyga, 10% Intravenous Solution — Panzyga is a 10% Ig formulation for intravenous (IV) administration
  Arms: Panzyga 10%
Other: Placebo — 4 mL/kg 0.9% w/v sodium chloride solution per single IV infusion
  Arms: Placebo

SUMMARY:
A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of Panzyga for Prevention of Major Infection in Patients with Hypogammaglobulinemia and Autoimmune or Rheumatic Conditions Receiving Treatment with B-cell Depletion Therapy

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria will be eligible to participate in the study:

1. Are ≥18 years of age at time of informed consent, have been diagnosed with a rheumatic or autoimmune condition, received their last BCDT dose within 3 months of Screening, and have the intention to receive BCDT during study participation. Note: Patients with the following indications are eligible: MS, RA, vasculitis/myositis, SLE, SS, IIM, MCTD, UCTD, myasthenia gravis, autoimmune encephalitis, CIDP, and neuromyelitis optica spectrum disorder). Other rheumatic and autoimmune conditions may also be acceptable with approval from the Medical Monitor.
2. Have hypogammaglobulinemia (IgG levels <5 g/L as confirmed by the central laboratory).
3. Are willing and able to provide voluntary written informed consent for participation in the study and to comply with all protocol requirements..
4. Are willing and able to comply with a highly effective contraception method during and for 30 days after the treatment period. Contraceptive use by men and women of childbearing potential should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from participation in the study:

1. Have a history of anaphylaxis or severe systemic response to immunoglobulin, blood, or plasma-derived products, or any Panzyga component
2. Have a current major infection at Screening or had >1 major infection within 6 months prior to Baseline
3. Have a history of thromboembolic events such as deep vein thrombosis, pulmonary embolism, myocardial infarction, ischemic stroke, transient ischemic attack, or peripheral artery disease (Fontaine IV) within 6 months prior to Baseline
4. Have a known IgA deficiency with antibodies to IgA
5. Have a known blood hyperviscosity or other hypercoagulable states
6. Have been diagnosed with primary immunodeficiency.
7. Have a severe liver disease, with signs of ascites or hepatic encephalopathy
8. Have a severe kidney disease (as defined by eGFR <30 mL/min/1.73 m2)
9. Have a body weight >140 kg
10. HIV infection at Screening (defined for the study as positive HIV NAT test or reactive HIV- 1/2 antigen/antibody immunoassay followed by positive HIV-1/HIV-2 antibody differentiation immunoassay)
11. Patients found to be chronic carriers of hepatitis B virus (HBV), defined by positive surface antigen (HBsAg), positive Hepatitis B core antibodies (HBcAb) and/or low HBV titers, who will not receive targeted antiviral therapy while participating in the study, and patients with active HBV, defined as high HBV titers.
12. Uncontrolled hepatitis C infection at Screening (defined for the study as positive HCV PCR).
13. Have received IgG treatment within 6 months prior to Screening or plan to receive IgG therapy, other than IMP, during the study
14. Are receiving or plan to receive immunosuppressive treatment (other than for underlying condition) or other forbidden medication during the entire study duration
15. Are participating or plan to participate in another study that is either blinded or involves an investigational medicinal product within 3 months prior to Baseline or during the course of this study. Participation in observational or open-label studies involving an approved product may be permitted after consultation with the Medical Monitor.
16. If female, are pregnant or lactating
17. Are likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem or poor mental development, in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Major Infections in Participants | 48 weeks
  Occurrence of at least one major infection or death in patients with or without primary infection prophylaxis with Panzyga during the treatment period. Each potential infection will be assessed by an Independent Adjudication Committee (IAC). Major infections will be defined as bacterial and/or viral infections, which are microbiologically documented or clinically documented requiring treatment with anti-infective, including those resulting in death, excluding confirmed cases of COVID-19.

SECONDARY OUTCOMES:
Time to Major Infections in Participants | 48 weeks
  Time to first major infection (as assessed by the IAC) during the treatment period or death. The secondary safety endpoints of this study include the incidence of adverse events and changes from baseline in physical examinations and clinical laboratory parameters.
Number of Participants Experiencing AEs | 48 weeks
  Incidents of AEs during the treatment period
Participants Experiencing Changes from Baseline in Physical Examinations, and Clinical Laboratory Parameters | 48 Weeks
  Changes from baseline in physical examination findings and clinical laboratory parameters will be assessed during the treatment period. Each parameter will be reported separately according to its unit of measure, such as body weight (kg), height (cm), body mass index (kg/m²), and individual laboratory values (e.g., hemoglobin [g/dL], serum creatinine [mg/dL]). Where applicable, related measurements (e.g., weight and height) will be combined to derive a single parameter, such as body mass index, to ensure consistent and interpretable results.

IPD SHARING:
Plan to Share IPD: No